CLINICAL TRIAL: NCT03307733
Title: Walking in Pregnancy (WiP) - a Social Networking Physical Activity Intervention for Pregnant Obese Women
Acronym: WiP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Hallam University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STH19365
Record Dates: First submitted 2017-08-23; First posted 2017-10-12 (Actual); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Maternal Obesity Complicating Pregnancy; Maternal Obesity Complicating Childbirth
MeSH Terms: interventions — Walking

STUDY DESIGN:
Intervention Model Description: Feasibility Randomized Control Trial
Masking Description: It is difficult to mask in these type of interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Control group received usual care plus a blinded Fitbit pedometer.
- Intervention (Active Comparator): Intervention group received a Fitbit pedometer with individualised physical activity targets and behaviour change techniques which were delivered via a closed Facebook group
  Interventions: Behavioral: walking and behavour change techniques

INTERVENTIONS:
Behavioral: walking and behavour change techniques — a Fitbit pedometer with individualised step targets and partaking in a closed Facebook group
  Arms: Intervention

SUMMARY:
A physical activity feasibility randomised control trial for pregnant, obese women.

DETAILED DESCRIPTION:
Overweight (defined as BMI ≥25kg/m2) and obesity (defined as BMI ≥30kg/m2) during pregnancy is becoming more common. Approximately 25-30% of women of childbearing age are obese and around 50% are overweight at the time of conception. Women who are either overweight or obese have a much higher risk of adverse pregnancy outcomes. For example, they are more likely to develop gestational diabetes, pregnancy-induced hypertension, pre-eclampsia, Caesarean section and other complications. Recent research suggests that overweight and obese pregnant women are less active than normal weight ( BMI≤ 25kg/m2) pregnant women and also that the level of physical activity decreases throughout pregnancy. The evidence also suggests that maintaining a good level of physical activity can reduce the risks of adverse pregnancy outcomes. A large study which looked at the most preferred types of physical activity identified that walking and swimming were the most preferred types of physical activity by pregnant women. Although there is an association between walking at a brisk pace and a reduced risk of gestational diabetes, there is no definitive conclusion on the effectiveness of walking interventions. The investigators are proposing this feasibility study in order to find out whether a walking intervention can be implemented during pregnancy in the obese population to reduce adverse pregnancy health outcomes. The current study will investigate whether a Fitibit Pedometer and a Social networking Site (Facebook) can be used to encourage pregnant, obese women to increase and maintain activity during pregnancy. The feasibility study will test the recruitment strategy, acceptability of the intervention design, randomisation acceptability, and timing of the intervention. Participants from both the control and the intervention will be purposefully selected to take part in focus group following the intervention in order to give feedback on the study. The investigators will be working with an Obstetrics & Gynaecology consultant at Jessop Wing, Hallamshire Hospital to help with the recruitment process and provide clinical advice. Women who are obese (BMI>30kg/m2) in their early pregnancy (12-14 weeks) will be recruited. Participants that consent to take part in the study will be given a Fitbit pedometer and enrolled in a closed Facebook group. Each participant will wear a Fitbit for a week in order to measure their baseline physical activity level. Thereafter, the participants in the intervention will be asked to gradually increase their physical activity level (they will be given a weekly step target)for 4 weeks in total. The Facebook component of the intervention will contain motivational and educational posts and rewarding messages about their progress. The control group will be asked to wear a Fitbit for 5 weeks and do their usual activities in total with a covered screen so as to not see the step count

ELIGIBILITY:
Inclusion Criteria:

* pregnant 11-14 weeks gestation
* BMI >30kg/m2
* No known risks or complications
* Able to walk

Exclusion Criteria:

* High risk of miscarriage

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — only women can be pregnant
Enrollment: 40 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
Recruitment | 5 weeks
  Recruitment rate will be calculated by simple descriptive statistics. (number of participants approached vs. number of participants that agree to take part)
Compliance | 5 weeks
  Compliance to the study procedures will be calculated by simple descriptive. statistics
Attrition | 5 weeks
  Drop out rate will be calculated by simple descriptive statistics.
Adherence rates | 5 weeks
  Adherence to Fitbit will be measured daily.

SECONDARY OUTCOMES:
Gestational Weight Gain | 5 weeks
  Women are recruited at 11-14 weeks gestation and after 5 weeks when they are at 20 weeks gestation the final assessments will be collected. Weight is measured in kilograms.
gestational diabetes status | 26 weeks
  Outcome of the gestational diabetes mellitus test at 26 weeks gestation.
Pregnancy and Birth outcomes | 9 months
  Preeclampsia ( Percentage figure of patients who developed preeclampsia during birth will be calculated from clinical notes).
C-section | 9 months
  Mode of Delivery ( Number of participants from each group who have a C-section will be calculated)
Birth weight | At delivery ( 9 months roughly)
  Weight of the baby at birth. This data will be collected from clinical notes.
Apgar score | At delivery ( 9 months roughly)
  5 minute Apgar Score. Score data will be collected from clinical notes.

IPD SHARING:
Plan to Share IPD: Undecided